CLINICAL TRIAL: NCT01455038
Title: Heart Rate Variability of Patients With Bipolar Disorder in Subsyndromal Depressive Phase
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Korean Health Technology R&D Project, Ministry of Health & Welfare (Unknown)
Responsible Party: Principal Investigator, Yeon-Ho Joo, Professor, Asan Medical Center
Other Study IDs: A090116
Record Dates: First submitted 2011-10-18; First posted 2011-10-19 (Estimated); Last update posted 2011-10-19 (Estimated); Status verified 2011-10

CONDITIONS: Bipolar Disorder; Subsyndromal Depressive Phase; Heart Rate Variability
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Control group: Healthy controls had no history of psychiatric disorder and had no psychiatric symptom when interviewed by a board-certified psychiatrist.
- Bipolar group: individual patient as being in subsyndromal depressive phase when the patient had a Montgomery-Åsberg depression rating scale score of 10 or less and Clinical Global Impression severity of 3 or less for last one month.

SUMMARY:
The purposes of this study were: (1) to compare heart rate variability between bipolar patients in subsyndromal depressive phase and healthy controls (2) to evaluate the relation between the severity of subsyndromal depressive symptoms and reduced heart rate variability.

ELIGIBILITY:
Inclusion Criteria:

1. Bipolar group:

   * DSM-IV bipolar disorder
   * Montgomery-Åsberg depression rating scale (MADRS) score for last one month : ≤ 10
   * Clinical Global Impression severity (CGI-S) for last one month : ≤ 3
2. Healthy controls group: Subjects had no history of psychiatric disorder and had no psychiatric symptom when interviewed by a board-certified psychiatrist.

Exclusion Criteria:

* Psychiatric disorder except bipolar disorder
* Neurological symptoms or signs
* History of head trauma
* History of cardiovascular diseases
* Any medication except psychiatric medication.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Thirty three (10 males, 23 females) patients in clinically remitted state diagnosed with bipolar disorder based on DSM-IV criteria were enrolled at one outpatient psychiatric clinic and 59 healthy controls (23 males, 36 females) from health promotion center in a university-affiliated general hospital. We defined an individual patient as being in subsyndromal depressive phase when the patient had a Montgomery-Åsberg depression rating scale (MADRS) score of 10 or less and Clinical Global Impression severity (CGI-S) of 3 or less for last one month. Healthy controls had no history of psychiatric disorder and had no psychiatric symptom when interviewed by a board-certified psychiatrist.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | at baseline
  Time domain - NN (normal-to-normal R-R interval), HRV index (total number of all NN/ the height of the histogram of all NN), SDNN (standard deviation of the NN), RMSSD (the root mean square of differences of successive NN), NN50 (Number of pairs of adjacent NN intervals differing by more than 50 ms in the entire recording) and pNN50(NN50/total number of all NN).
  Frequency domain - TP (The variance of NN intervals over the temporal segment), VLF(Power in very low frequency range; <0.04 Hz), LF(Power in low frequency range; 0.04~0.15 Hz), HF(Power in high frequency range; 0.15~0.4 Hz)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea